CLINICAL TRIAL: NCT00711360
Title: Monitoring of Fluid Status in Heart Failure Patients by Intrathoracic Impedance Measurement
Brief Title: Monitoring of Fluid Status in Heart Failure Patients by Intrathoracic Impedance Measurement (HomeCARE II)
Acronym: HomeCARE II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TA083; There is no secondary ID
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure; Arrhythmias, Cardiac
Keywords: heart failure; implantable cardioverter-defibrillator; intrathoracic impedance; cardiac resynchronization therapy; home monitoring
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intrathoracic impedance measurement — Intrathoracic impedance measurement by cardiac resynchronization therapy (CRT) devices and implantable cardioverter defibrillators (ICDs) (Lumax 540)

SUMMARY:
The new BIOTRONIK implantable cardioverter defibrillator (ICD) family Lumax 540 is capable of measuring the intrathoracic impedance on a daily basis and transmission of impedance trend data via the Home Monitoring technology. In future, this will allow for automatic early detection of imminent decompensation at a presymptomatic stage and immediate initialization of clinical meaningful therapeutic interventions preventing heart failure related hospitalizations. The aim of this investigation is to record long-term impedance trends in heart failure patients with and without heart failure related events (hospitalizations due to acute decompensation) in order to develop algorithms for device-based early detection and warning of HF deterioration accompanied by pulmonary congestion.

DETAILED DESCRIPTION:
The new BIOTRONIK implantable cardioverter defibrillator (ICD) family Lumax 540 is capable of measuring the intrathoracic impedance on a daily basis and transmission of impedance trend data via the Home Monitoring technology. In future, this will allow for automatic early detection of imminent decompensation at a presymptomatic stage and immediate initialization of clinical meaningful therapeutic interventions preventing heart failure related hospitalizations. The aim of this investigation is to record long-term impedance trends in heart failure patients with and without heart failure related events (hospitalizations due to acute decompensation) in order to develop algorithms for device-based early detection and warning of HF deterioration accompanied by pulmonary congestion.

Lumax is the name of a family of implantable ICDs. The primary objective of the therapy is the prevention of sudden cardiac death. The aim is to automatically detect and terminate cardiac arrest caused by ventricular tachyarrhythmia. All major therapeutical approaches from the field of cardiology and electrophysiology are contained within the Lumax family.

Furthermore, the device is capable of treating bradycardia arrhythmias and congestive heart failure. Congestive heart failure is treated with cardiac resynchronization therapy with multisite ventricular pacing known as cardiac resynchronization therapy (CRT).

The integrated Home Monitoring component can provide information about occurring rhythm disturbances and delivered therapies close to real time as well as by intracardiac electrogram (IEGM) Online HD®. Furthermore, statistical data about the patient's condition as well as information about the integrity status of the implant itself are sent.

The implantation of an ICD is a symptomatic therapy with the following objectives:

* Termination of spontaneous ventricular fibrillation (VF) through shock delivery
* Termination of spontaneous ventricular tachycardia (VT) by means of antitachycardia pacing (ATP); in case of ineffective ATP or hemodynamically not tolerated VT with shock delivery
* Cardiac resynchronization by multisite ventricular pacing (triple-chamber implant)
* Compensation of bradycardia through ventricular (single-chamber implant) or atrioventricular sequential pacing (dual- and triple-chamber implant)

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for 1-, 2- or 3-chamber ICD implantation according to current guidelines or patient already implanted with a Lumax 540 device or successor
* NYHA-class II to IV
* LVEF lower or equal to 35%
* Patient accepts Home Monitoring concept and has sufficient GSM/GPRS net coverage
* Increased risk for HF-related hospitalization according to pre-defined criteria
* Patient information
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Contraindication for ICD implantation
* Post HTX or actively listed for HTX
* Cardiac surgery within the previous 3 months or planned at time of inclusion
* Acute coronary syndrome within the previous 3 months
* Chronic renal dialysis
* Pregnant or breast-feeding women
* Limited contractual capability
* Participation in another study
* Anticipated non-compliance with the follow-up scheme
* Life expectancy not longer than 1.5 years due to a non-cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Long-term impedance trends in patients with clinically relevant heart failure events, to support the development of impedance based detection algorithms. A posterior assessment of sensitivity and false alarm rate of the detection algorithms. | Study will last until 35 heart failure events are collected

SECONDARY OUTCOMES:
Further improvement of the Heart Failure Monitor based on collected data | The same as for primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Maier, PD Dr. med., Study Chair — Medizinische Klinik und Poliklinik I Universitätsklinikum Würzburg, Germany
Locations (28):
- Germany (24):
  - RWTH Medizinische Klinik I Aachen, Aachen
  - Klinikum Aschaffenburg, Aschaffenburg
  - Kerckhoff-Klinik GmbH Bad Nauheim, Bad Nauheim
  - Herz- und Gefäss-Klinik GmbH Bad Neustadt, Bad Neustadt A. D. Saale
  - HDZ Bad Oeynhausen NRW, Bad Oeynhausen
  - Universitätsklinikum Benjamin Franklin, Berlin
  - Berufsgenossenschaftliche Kliniken Bergmannsheil Universität Bochum, Bochum
  - Kliniken Erlabrunn gGmbH, Breitenbrunn
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Ernst-Moritz-Arndt Universität Greifswald, Greifswald
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Städtische Kliniken Neuss -Lukaskrankenhaus- GmbH, Neuss
  - Marienhospital Osnabrück GmbH, Osnabrück
  - Marienkrankenhaus Papenburg-Aschendorf GmbH, Papenburg
  - St. Elisabeth Klinik Saarlouis, Saarlouis
  - Krankenhaus der Evangelischen Diakonissenanstalt, Speyer
  - Universitätsklinikum Tübingen, Tübingen
  - Kliniken Villingen, Villingen
  - Universitätsklinikum Würzburg, Würzburg
- Spain (3):
  - Hospital General Yagüe, Burgos
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital General universitario Valencia, Valencia
- Cardio Centro Ticino, Lugano, Switzerland

REFERENCES:
- [Derived] Maier SKG, Paule S, Jung W, Koller M, Ventura R, Quesada A, Bordachar P, Garcia-Fernandez FJ, Schumacher B, Lobitz N, Takizawa K, Ando K, Adachi K, Shoda M. Evaluation of thoracic impedance trends for implant-based remote monitoring in heart failure patients - Results from the (J-)HomeCARE-II Study. J Electrocardiol. 2019 Mar-Apr;53:100-108. doi: 10.1016/j.jelectrocard.2019.01.004. Epub 2019 Jan 25. PMID 30739055